CLINICAL TRIAL: NCT02191969
Title: The Impact of a Physical Activity Intervention in Older Patients Undergoing Adjuvant Chemotherapy for Colorectal Cancer: a Randomized, Controlled Trial
Brief Title: Physical Activity Intervention for Older Patients During Chemotherapy for Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: LCCC Geriatric Oncology Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1324
Record Dates: First submitted 2014-06-17; First posted 2014-07-16 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer; Fatigue
Keywords: Chemotherapy; Adjuvant Chemotherapy; Cancer Therapy; Fatigue; Physical Activity; Physical Function; Tiredness; Colon Cancer; Rectal Cancer; Walk With Ease; Colorectal Cancer; Geriatric Assessment; Geriatric; Elderly
MeSH Terms: conditions — Colorectal Neoplasms; Fatigue; Motor Activity; Colonic Neoplasms; Rectal Neoplasms | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This group will be receiving adjuvant chemotherapy for colorectal cancer. They will not participate in the Walk With Ease program. They will be followed up using standard of care.
- Intervention (Experimental): This group will be receiving adjuvant chemotherapy for colorectal cancer. They will participate in the Walk With Ease (WWE) program during the course of their chemotherapy treatment. They will be requested to initiate the WWE starting on Day 1 of adjuvant chemotherapy. Participants are asked to walk at a safe and comfortable pace, increasing their minutes per day at a rate they can sustain, with the ultimate goal of 30 minutes/day for at least 5 days/week. They are asked to maintain a daily walking log that is provided to them, entering total minutes per day.
  Participants will be asked to do the walking program independently (self-directed, not in a formal group with an instructor) throughout chemotherapy.
  Interventions: Behavioral: Walk With Ease

INTERVENTIONS:
Behavioral: Walk With Ease — A self-directed walking intervention developed by the Arthritis Foundation. The intervention is a workbook that coaches participants through walking regularly at a safe, comfortable pace with the ultimate goal of walking at least 30 minutes a day five days a week.
  Other Names: WWE
  Arms: Intervention

SUMMARY:
This study will see if patient who undergo a physical activity intervention called Walk With Ease report experiencing less fatigue and a higher quality of life during chemotherapy for colorectal cancer than those who do not participate in this intervention.

DETAILED DESCRIPTION:
The primary purpose of this multicenter, randomized controlled study is to evaluate the impact of a physical activity program on fatigue in older patients (≥60 years) undergoing adjuvant chemotherapy for colorectal cancer. The investigators also plan to evaluate physical function and quality of life as secondary objectives. The investigators' hypotheses are that people who undergo the physical activity intervention compared to those who do not, will: 1) report less fatigue, 2) report higher health related quality of life, and 3) have less decline in physical function. Additionally, The investigators will characterize ≥grade 3 adjuvant chemotherapy associated toxicities in this older population, and describe the changes reported in fatigue, physical function, and HRQOL over the course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ Age 60 years (no upper age limit)
* Diagnosis of stage II-III colon or rectal cancer planned for treatment with adjuvant chemotherapy scheduled as part of standard treatment
* Able to read English (required for CGA and other surveys administered)
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Signed, IRB-approved written informed consent

Exclusion Criteria:

* Other active, invasive malignancy requiring ongoing therapy or expected to require systemic therapy
* Already walking or engaging in other physical activity >120 minutes per week as documented via subject self-report
* Unable to walk or engage in moderate-intensity physical activity
* One or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
To measure the change in fatigue after three months between the intervention and control arm | Three Months
  The investigators will compare the change in fatigue from baseline to 3 months between Intervention and Control arms as measured via PROMIS®-Fatigue.

SECONDARY OUTCOMES:
To measure changes in physical function at baseline between the intervention and control groups. | 4 to 24 weeks
  To evaluate the following measures at baseline, 3 months, and after completion of chemotherapy and compare changes in these measures over time between Intervention and Control arms.
  • Physical function as measured by PROMIS-PF and SPPB
To measure adherence to the physical activity intervention | One Year
  To report on the adherence of the physical activity intervention as measured through self-reported minutes of walking per days and walking minutes per week in the group randomized to the Intervention arm
To measure the difference in p16INK4a levels before and after chemotherapy in the control and intervention groups | One Year
  The investigators will comparee the change in p16INK4a and muscle mass measurements pre/post adjuvant chemotherapy between Intervention and Control groups
To measure the change in muscle mass measurements before and after chemotherapy between the intervention and control arms | One Year
  The investigators will compare the change in p16INK4a and muscle mass measurements pre/post adjuvant chemotherapy between Intervention and Control groups
To measure the association of p16INK4a and muscle mass with any differences in fatigue o physical function or QOL during chemotherapy | Six months
  To explore the association of baseline measurements of p16INK4a and muscle mass with changes in fatigue, physical function, and health related quality of life during adjuvant chemotherapy.
To measure changes in Quality of Life at baseline between the intervention and control groups. | 4 to 24 weeks
  To evaluate the following measures at baseline, 3 months, and after completion of chemotherapy and compare changes in these measures over time between Intervention and Control arms.
  Quality of life as measured by FACT-FCSI and PROMIS-PI
To measure changes in ADLs at baseline between the intervention and control groups. | 4 to 24 weeks
  To evaluate the following measures at baseline, 3 months, and after completion of chemotherapy and compare changes in these measures over time between Intervention and Control arms.
  ADLs per CGA
To measure changes in Instrumental Activities of Daily Living at baseline between the intervention and control groups. | 4 to 24 weeks
  To evaluate the following measures at baseline, 3 months, and after completion of chemotherapy and compare changes in these measures over time between Intervention and Control arms.
  IADLs per CGA
To measure changes in Self-Efficacy at baseline between the intervention and control groups. | 4 to 24 weeks
  To evaluate the following measures at baseline, 3 months, and after completion of chemotherapy and compare changes in these measures over time between Intervention and Control arms.
  Self-efficacy and attitudes as measured by PSEFSM and OEE

CONTACTS AND LOCATIONS:
Overall Officials: Hy Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Williams GR, Nyrop KA, Deal AM, Muss HB, Sanoff HK. Self-directed physical activity intervention in older adults undergoing adjuvant chemotherapy for colorectal cancer: Design of a randomized controlled trial. Contemp Clin Trials. 2015 May;42:90-7. doi: 10.1016/j.cct.2015.03.008. Epub 2015 Mar 28. PMID 25827253
- See also: The Geriatric Oncology Research Program at UNC — https://unclineberger.org/patientcare/programs/geriatric